CLINICAL TRIAL: NCT05116826
Title: An Open-label, Phase 1, Multiple-dose Study to Evaluate the Pharmacokinetics of Nitazoxanide 500 mg Twice Daily for 7 Days in Adult Subjects With Moderate and Severe Hepatic Impairment and Adult Healthy Control Subjects
Brief Title: Nitazoxanide Pharmacokinetic Parameters in Hepatic Impaired Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NTZ-121-1
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Moderate Hepatic Impairment; Severe Hepatic Impairment; Liver Diseases
Keywords: Pharmacokinetics; Healthy Volunteer; Liver Disease; Hepatic Impairment; Antiparasitic; Antiprotozoal
MeSH Terms: conditions — Liver Diseases | interventions — nitazoxanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Control Match (Normal hepatic function) (Experimental): NTZ 500 mg twice a day for 7 days
  Interventions: Drug: Nitazoxanide
- Moderate Child-Pugh B (Moderate hepatic impairment) (Experimental): NTZ 500 mg twice a day for 7 days
  Interventions: Drug: Nitazoxanide
- Severe Child-Pugh C (Severe hepatic impairment) (Experimental): NTZ 500 mg twice a day for 7 days
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — 500 mg Twice Daily for 7 days
  Other Names: NTZ

SUMMARY:
This study is being conducted to evaluate the major Nitazoxanide (NTZ) active metabolite in adult participants with hepatic impairment and healthy adults.

DETAILED DESCRIPTION:
This study is being conducted to assess the effect of hepatic impairment on the pharmacokinetics of the major Nitazoxanide active metabolite in hepatic impaired (moderate and severe according to Child-Pugh categories) and healthy control adults following repeated oral dose administration of NTZ 500 mg twice a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 75 years of age, inclusive;
2. With a minimum body weight of 50 kg and within a BMI range of 18.0 to 40.0 kg/m^2, inclusive;
3. Females participating in this study must be of non-childbearing potential or must be using highly effective contraception for the full duration of the study;
4. Negative human immunodeficiency virus antibody screens at Screening;
5. Matched to participants with moderate and/or severe hepatic impairment in age (± 10 years), BMI (± 20 percentage) and sex;
6. Participants who have chronic (≥ 6 months) moderate or severe hepatic insufficiency (of any etiology) that has been clinically stable (no acute episodes of illness due to deterioration in hepatic function) for at least 1 month prior to Screening and must also remain stable throughout the Screening period.

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

1. A positive alcohol test result at Check-In Visit;
2. A history of alcohol abuse in the prior 2 years;
3. Positive urine screen for drugs of abuse at Screening or Check-In;
4. Strenuous exercise within 72 hours prior to Check-In Visit;
5. Blood donation or loss of blood (excluding volume drawn at screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing;
6. History of a major surgical procedure within 30 days prior to Screening;
7. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed. Bariatric surgery will not be allowed;
8. Presence or history of malignancy within the prior 3 years, with the exception of treated basal cell or squamous cell carcinoma;
9. Poor peripheral venous access;
10. Receipt of blood products within 2 months prior to Check-In Visit;
11. Significant history or clinical manifestation of any metabolic (including thyroid), allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal (GI), neurological, or psychiatric disorder;
12. Positive serologic test for hepatitis B surface antigen or for hepatitis C virus antibody at Screening;
13. Frequent headaches (> twice a month) and/or migraines, recurrent nausea and/or vomiting, diarrhea;
14. Participants with symptomatic hypotension at Screening, whatever the decrease of blood pressure, or asymptomatic postural hypotension;
15. History of unstable diabetes mellitus;
16. Participants who have a transjugular intrahepatic portosystemic shunt and/or have undergone portacaval shunting;
17. Participant has shown evidence of hepatorenal syndrome or has creatinine clearance ≤ 60 mL/min;
18. Participants has required treatment for GI bleeding within the 6 months prior to Check-In Visit;
19. Recent history of paracentesis (< 1 months prior to Check-In Visit);
20. Participants with Wilson's disease, alpha-1 antitrypsin deficiency, glycogen storage diseases, or galactosemia;
21. Participants with anemia secondary to hepatic disease, unless hemoglobin is ≥ 8.5 g/dL and anemia symptoms are not clinically significant. Participants must have ≥ 30,000 platelets at screening and at Check-In Visit.

Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) from time zero to 12h (AUC0-12) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 hours post dose
  In participants with moderate and severe hepatic impairment compared to healthy volunteers
AUC from time zero to the time of the last quantifiable concentration (AUC0-t) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 hours post dose
  In participants with moderate and severe hepatic impairment compared to healthy volunteers
Maximum observed plasma concentration (Cmax), | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 hours post dose
  In participants with moderate and severe hepatic impairment compared to healthy volunteers

SECONDARY OUTCOMES:
Plasma pharmacokinetics: time of the maximum observed plasma concentration (Tmax), apparent plasma terminal elimination half life (t1/2), AUC from time zero to infinity (AUC0-∞), trough concentration (Ctrough) and percentage of extrapolated (%AUCextrap) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 hours post dose
  For NTZ and its major active metabolite
Plasma pharmacokinetics: Tmax, AUC0-12, AUC0-t, AUC0-∞, Cmax, t1/2, %AUCextrap and Ctrough. | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 hours post dose
  For the NTZ major active metabolite
Urine pharmacokinetics: amount of drug excreted (Ae), cumulative amount of drug excreted (Ae0-t), and renal clearance (CLR) | Day-1: pre-dose, Day 1: 0-4 h, 4-8 h, 8-12, 12-24 h post-dose; Day 7: 0-4 h, 4-8 h, 8-12 h, 12-24 h, 24-48 h post-dose
  For the NTZ major active metabolites
Plasma and urine pharmacokinetics: After the single oral administration of NTZ 500 mg: Cmax, AUC0-12, AUC0-t, AUC0-∞ , Tmax, t1/2, %AUCextrap, Ae0-∞, Ae0-t and CLR. | Plasma:Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10, 12 h post dose Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24; and 48 h post dose Urine:Day-1: pre-dose, Day 1: 24 hours urine collection post-dose; Day 7: 48 hours urine collection
  For the NTZ major active metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Carol Addy, MD, Study Director — Genfit
Locations (2):
- United States (2):
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No